CLINICAL TRIAL: NCT05429905
Title: Dual Anti-CD22/CD19 Chimeric Antigen Receptor-directed T Cells (CART2219.1) for Relapsed Refractory B-Lineage Leukaemia
Status: Unknown | Phase: Phase 1 / Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: KK Women's and Children's Hospital (Other Government)
Collaborators: Singapore General Hospital (Other); National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: CART2219-1.0
Record Dates: First submitted 2021-12-16; First posted 2022-06-23 (Actual); Last update posted 2023-03-09 (Actual); Status verified 2023-03

CONDITIONS: Lymphoblastic Leukemia; Lymphoblastic Leukemia, Acute, Childhood; Lymphoblastic Leukemia in Children; Lymphoblastic Leukemia, Acute Adult; CAR
Keywords: CAR T-cell therapy; B-ALL; Relapsed/ Refractory
MeSH Terms: conditions — Precursor Cell Lymphoblastic Leukemia-Lymphoma | interventions — Clinical Trials, Phase I as Topic; Clinical Trials, Phase II as Topic

STUDY DESIGN:
Intervention Model Description: Phase 1 run-in will be conducted to determine the recommended phase II dose(s) (RP2D) for adult and paediatric patients in independent dose escalation cohorts.
  Phase II will enrol patients in 2 concurrent cohorts at the R2PD.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1 (Dose-escalation) (Experimental): Dose-finding and dose expansion cohort for intravenous autologous anti-CD22/CD19 CAR-T using a relapsed refractory B-ALL cohort.
  Interventions: Biological: Phase I
- Cohort 2 (High MRD) (Experimental): Patients with B-ALL with high MRD after induction therapy or after consolidation therapy in replacement of stem cell transplant
  Interventions: Biological: Phase II
- Cohort 3 (Extramedullary ALL) (Experimental): Patients with testicular or central nervous system B-ALL in replacement of radiation
  Interventions: Biological: Phase II

INTERVENTIONS:
Biological: Phase I — * Dose level 0: CAR+CD3+ 0.4 x 10e6/kg (de-escalation dose)
  * Dose level 1: CAR+CD3+ 1 x 10e6/kg (starting dose)
  * Dose level 2: CAR+CD3+ 2.5 x 10e6/kg.
  Dose-escalations for adults and paediatrics will be performed in 2 independent strata for determination of RP2D.
  Arms: Cohort 1 (Dose-escalation)
Biological: Phase II — RP2D will be determined in Phase I
  Arms: Cohort 2 (High MRD); Cohort 3 (Extramedullary ALL)

SUMMARY:
The purpose of this study is to deliver dual-targeting CAR-T cell therapy (CART 2219.1) as a salvage treatment to patients with relapsed/refractory B-lineage leukaemia in place of stem cell transplant or irradiation.

ELIGIBILITY:
Inclusion Criteria:

All Cohorts:

* Age 2 to 75 years
* Absolute blood CD3+ T cell count ≥100/μl
* ECOG performance score of ≤2 if >16 years old, or Lansky performance score of >50 if ≤16 years old at screening
* Patients and/or parents must give their written informed consent/assent.
* Patients have relapsed/refractory B-lineage acute lymphoblastic leukaemia, includes persistent minimal residual disease (MRD)

Cohort 1 (Phase I): Relapsed/Refractory B-ALL

* Patients must have relapsed/refractory (r/r) B-lineage ALL meeting one of the following disease-specific criteria:

  * Patients with r/r ALL with >5% blasts in BM (M2 or M3) after at least one standard chemotherapy and one salvage regimen who are ineligible for allogeneic stem cell transplant (alloSCT) or have refractory disease activity (e.g. persistent MRD in bone marrow) precluding alloSCT, or
  * Patients with Ph+ ALL if they are intolerant to tyrosine kinase inhibitor (TKI) therapy, or if they have r/r disease after treatment including TKI, or
  * Patients who have relapsed post-allogeneic HSCT and are at least 100 days post-transplant, with no evidence of active GVHD, > 6 weeks post donor lymphocyte infusion (DLI) and no longer taking immunosuppressive agents for at least 30 days prior to enrolment.
  * Patients who have relapsed after prior CAR-T therapy who are not eligible for stem cell transplant and have < 5% circulating CAR-T prior to apheresis
* Patients with refractory/relapsed combined extramedullary ALL are eligible. This includes patients with combined CNS-2 (<5 WBC/μl CSF, with blasts on cytospin) or CNS-3 (>5 WBC/ul CSF, with blasts on cytospin) disease and patients with combined testicular relapse.

Cohort 2 (Phase II): B-ALL with persistent MRD (High Risk B-ALL)

• Patients must have persistent MRD >0.1% blasts after frontline induction chemotherapy or >0.01% blasts after consolidation therapy.

Cohort 3 (Phase II): Relapsed/Refractory Extramedullary B-ALL

* Patients with testicular leukaemia confirmed on biopsy
* Patients with CNS-3 B-ALL or Leptomeningeal disease
* Patients with combined bone marrow and extramedullary relapse (as defined in Cohort 1) are eligible.

Exclusion Criteria:

All Cohorts:

* Blasts are negative for both CD22 and CD19 on flow cytometry or immunohistochemistry, defined as < 10% of blasts staining positive for CD22 and CD19 respectively [IBFM 2016 Consensus Guidelines].
* Current autoimmune disease, or history of autoimmune disease with potential CNS involvement
* Active clinically significant CNS dysfunction (including but not limited to uncontrolled seizure disorders, cerebrovascular ischemia or hemorrhage, dementia, paralysis)
* History of an additional malignancy other than non-melanoma skin cancer or carcinoma in situ unless disease free for ≥3 years.
* Pulmonary function: Patients with pre-existing severe lung disease (FEV1 or FVC < 65%) or an oxygen requirement of >28% O2 supplementation or active pulmonary infiltrates on chest X-ray at the time scheduled for T cell infusion
* Cardiac function: Fractional shortening <28% or left ventricular ejection fraction <50% by echocardiography
* Renal function: Creatinine clearance <50 mL/min/1.73 m2
* Liver function: Patients with a serum bilirubin >3 times upper limit of normal or an AST or ALT > 5 times upper limit of normal, unless due to leukemic liver infiltration in the estimation of the investigator
* Rapidly progressive disease that in the estimation of the investigator would compromise ability to complete study therapy
* Active Hepatitis B (HBsAg positive) or Hepatitis C (PCR positive), or known infection with human immunodeficiency virus (HIV)
* Pregnant or nursing (lactating) women
* In relation to prior therapy:

  * Use of immunotherapy, cell-based or other investigational treatment within 30 days of CAR-T infusion

Ages: 2 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2022-07-18 (Actual); Primary Completion 2024-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Recommended Phase II Dose (Phase I, Cohort 1) | 30 days
  The RP2D will be the dose level at which < 1 DLT in 3 patients or < 2 DLT in 6 patients is observed in both the adult and paediatric dose escalation stratas.
Number of patients with dose-limiting toxicities (Phase I, Cohort 1) | 30 days
  To be DLTs, adverse events must be suspected to be secondary to CAR-T cell infusion, occur during the first 30 days after infusion and meet at least one of the following criteria:
  1. Grade ≥ 3 non-hematologic toxicities, with the following exceptions:
     * Laboratory abnormalities without associated symptomatology or clinical consequence that resolve in less than 7 days;
     * Grade ≤ 2 cytokine release syndrome;
     * Grade 3 cytokine release syndrome that improves to grade ≤ 2 within 3 days of intervention;
     * Grade 3 neurotoxicity that resolves to grade 2 or less within 3 days.
     * Laboratory abnormalities compatible with tumor lysis syndrome;
  2. Grade ≥ 4 hematologic toxicities that persist at a grade ≥ 3 for >21 days.
  Cytokine release syndrome and immune-effector cell associated neurotoxicity syndrome (ICANS) are graded according to ASTCT consensus grading. Adverse events are graded according to CTCAE version 5.0.
12-month Leukaemia Free Survival (Phase II, Cohort 2 and 3) | 12 months
  Survival with Marrow MRD <0.01% by flow cytometry

SECONDARY OUTCOMES:
Overall Survival Rate (OS) | 12 months
  Percentage of patients in the study who are alive 12 months after CAR-T infusion.
Overall Response Rate (ORR) | 3 months
  Percentage of patients in the study who have a partial or complete response to the treatment within 3 months.
Duration of Response (DOR) | Up to 24 months
  Duration of complete remission (CR or CR with partial/incomplete haematological recovery)
Duration of CAR-T persistence | Up to 24 months
  Duration of measurable CAR-T above detection limits in peripheral blood and/or marrow

CONTACTS AND LOCATIONS:
Overall Officials: Michaela Seng, MD, Principal Investigator — KK Women's and Children's Hospital, BMTCT; Wing Hang Leung, MD PhD, Study Chair — KK Women's and Children's Hospital, BMTCT
Locations (1):
- KK Women's and Children's hospital, Singapore, Singapore

IPD SHARING:
Plan to Share IPD: Undecided